CLINICAL TRIAL: NCT07197281
Title: Correlation Between Perfusion Index Ratio and End Diastolic Velocity Ratio After Supraclavicular Brachial Plexus Block as an Early Predictor of Successful Block in Superficialization Surgery of the Upper Limb
Brief Title: Perfusion Index and End Diastolic Velocity Ratios as Predictors of Supraclavicular Block Success in Vascular Access Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abubakr Ali, resident at the Anesthesia, Intensive Care, and Pain Management department, Assiut University
Other Study IDs: PI and EDV as Predictors
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: End Diastolic Velocity; Perfusion Index
Keywords: End Diastolic Velocity; brachial plexus block; Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients scheduled for elective superficialization surgery of the upper limb: Participants are adult patients aged 18-65 years, both male and female, classified as ASA II-VI, and scheduled for elective superficialization procedures (mainly AV fistula superficialization).

SUMMARY:
This is a prospective observational study investigating the correlation between Perfusion Index (PI) ratio and End Diastolic Velocity (EDV) ratio as early predictors of successful supraclavicular brachial plexus block (SCBPB) in patients undergoing superficialization surgery of the upper limb.

DETAILED DESCRIPTION:
Regional anesthesia is fundamental for upper limb surgeries, with SCBPB providing dense anesthesia. However, early confirmation of successful block performance remains challenging. Traditional clinical methods (sensory/motor testing) are subjective and delayed. This study proposes using objective, noninvasive indices - PI (evaluated via pulse oximetry) and EDV (measured by Doppler ultrasound) - to determine their accuracy in detecting sympathetic blockade shortly after SCBPB. Early and reliable detection of block success is particularly important in superficialization surgeries such as arteriovenous fistula (AVF) superficialization in patients with compromised vascular status. The results are expected to enhance anesthesia practice by providing quantitative, reproducible, and rapid assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years

Both genders

ASA II-VI classification

Undergoing elective upper limb superficialization surgery (e.g., AVF superficialization)

Provided written informed consent

Exclusion Criteria:

* Patient refusal

Coagulopathy or bleeding disorders

Local infection at injection site

Allergy to local anesthetics

Use of vasopressors or beta-blockers

Severe peripheral vascular disease

Morbid obesity (BMI > 35)

Severe neurological or psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are adult patients aged 18-65 years, both male and female, classified as ASA II-VI, and scheduled for elective superficialization procedures (mainly AV fistula superficialization). Patients must be capable of understanding and signing informed consent. Excluded are patients with contraindications to nerve block such as coagulopathy, local infection, allergy to local anesthetics, severe vascular disease, morbid obesity (BMI >35), severe neurological or psychiatric impairment, or those taking vasopressors or beta-blockers that could alter vascular reactivity.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Perfusion Index ratio | 15 minutes
  Change in Perfusion Index ratio at 15 minutes after supraclavicular brachial plexus block in predicting successful block
Change in End Diastolic Velocity ratio | 15 minutes
  Change in End Diastolic Velocity ratio at 15 minutes after supraclavicular brachial plexus block in predicting successful block

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelnasser A, Abdelhamid B, Elsonbaty A, Hasanin A, Rady A. Predicting successful supraclavicular brachial plexus block using pulse oximeter perfusion index. Br J Anaesth. 2017 Aug 1;119(2):276-280. doi: 10.1093/bja/aex166. PMID 28854539